CLINICAL TRIAL: NCT02732821
Title: Observational Study of the Efficacy and Outcomes of Gastric Peroral Endoscopic Myotomy (G-POEM) for Treatment of Refractory Gastroparesis
Brief Title: G-POEM for Treatment of Refractory Gastroparesis
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00066924
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Gastroparesis; Idiopathic Gastroparesis; Gastroparesis Postoperative
Keywords: Gastroparesis; G-POEM; Gastric Per Oral Endoscopic Myotomy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric Per Oral Endoscopic Myotomy: All patients presenting with Gastroparesis will undergo Per oral endoscopic gastric myotomy
  Interventions: Procedure: Gastric Per Oral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Gastric Per Oral Endoscopic Myotomy — Patients will receive Per Oral Endoscopic Gastric Myotomy for Gastroparesis.

SUMMARY:
This study is performed to assess the efficacy and outcomes of Gastric Per Oral Endoscopic Myotomy "G-POEM" in patients presenting with gastroparesis.

DETAILED DESCRIPTION:
Gastroparesis is a chronic digestive disorder best defined as severe nausea, vomiting, bloating, and abdominal pain in the setting of objectively delayed gastric emptying without mechanical gastric outlet obstruction. The most common etiology is idiopathic. Some of the identifiable etiologies include diabetes and post-surgical.

Endoscopic techniques to reduce pyloric tone mainly consisted of Botulinum toxin injection but failed to demonstrate significant symptom improvement compared to placebo. Another endoscopic method was transpyloric stenting which yielded symptomatic relief but is prone to stent migration and therefore is unlikely to provide a viable long term solution.

Surgical pyloroplasty has shown to be effective in reducing gastroparesis symptoms, but is associated with a risk of leakage and potential further narrowing of gastric outlet. It also carried all the risks of general anesthesia and requires advanced laparoscopic suturing skills. Therefore, the development of a less invasive reliable method of improving gastric emptying is highly desirable.

An endoscopic submucosal myotomy technique may be applied to divide the pyloric sphincter without surgical access. Such endoscopic technique may provide the benefits of a natural orifice procedure, and improve gastric emptying in gastroparetic patients. Gastric Per-Oral Endoscopic Myotomy (G-POEM) is feasible and can be performed by using techniques similar to those of esophageal per-oral endoscopic myotomy. Endoscopists who are experienced in esophageal per-oral endoscopic myotomy should be able to perform G-POEM because both use similar techniques, principles, and equipment.

The investigators theorize that a subset of patients with refractory gastroparesis, diabetic gastroparesis or post-surgical gastroparesis, may respond to endoscopic pyloromyotomy.

ELIGIBILITY:
Inclusion Criteria:

• Adult patient age greater than 18 years old who are undergoing a standard-of-care G-POEM procedure.

Exclusion Criteria:

* Previous surgery of the esophagus or stomach which has resulted in a resection of the antrum and pylorus
* Known active gastroesophageal malignancy
* Prior surgical or laparoscopic pyloromyotomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who initially approach the study team from outside the institution (e.g. responding to the clinicaltrials.gov listing) or patients seen in the gastroenterology clinic.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of the G-POEM | Up to 1 year
  Improvement in patients symptoms as evaluated by the Gastroparesis Cardinal Symptom Index (GCSI) at 1 month, 3 months, 6 months and 1 year.
  The GCSI consists of three sub-scales: nausea/vomiting (three items), post-prandial fullness/early satiety (four items) and bloating (two items). Each item is rated on a Likert scale ranging from 0 (none) to 5 (very severe). Subscales are the average of different sets of items and are reported as a number between 0 to 5.
  Efficacy will be defined as a decrease in the GCSI score average below 2.

SECONDARY OUTCOMES:
Patient symptom improvement | Up to 1 year
  Improvement in patients symptoms will be assessed using symptom severity score at 1 month, 3 months, 6 months and 1 year.
  Symptoms will be recorded with a standardized gastroesophageal symptom assessment tool using a scale of 0-4 with higher ordinal values representing the greater frequency of symptoms for nausea, vomiting, bloating, abdominal pain, Gastroesophageal Reflux Disease (GERD) symptoms.
Delayed gastric emptying using a Gastric emptying study | 3 months
  Assess efficacy of the G-POEM in the treatment of gastroparesis using gastric emptying study to assess delayed gastric emptying by measuring the average percentage of 4-hour gastric retention of a solid meal.
Imapct of the G-POEM on patients' Quality of life | Up to 1 year
  Improvement in patient's quality of life as reflected by Short Form 36 questionnaire at 1 month, 3 months, 6 months and 1 year after the procedure.
  The SF-36 general health questionnaire consists of 36 questions evaluating the patient's perception of their quality of life (QoL) in the following eight subscales: physical functioning (PF), role limitations due to physical problems (RP), role limitations due to emotional problems (RE), energy/fatigue (EF), emotional well-being (EW), social functioning (SF), bodily pain (BP) and general health (GH). Subscale scores range from 0 to 100, with 100 being the best and 0 being the worst quality of life.
Efficacy of the G-POEM | 1 year
  Improvement in patients symptoms as evaluated by gastroparesis specific symptom assessment (PAGI-SYM questionnaire).
  PAGI-SYM is a 20-item self-reported questionnaire which evaluates the symptom severity of upper gastrointestinal disorders across six subscales (nausea/vomiting, fullness/early satiety, bloating, upper abdominal pain, lower abdominal pain and heartburn/regurgitation). These are summarized by individual subscale scores and a total score. Each item is rated on a Likert scale ranging from 0 (none) to 5 (very severe). Subscales are the average of different sets of items and are reported as a number between 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vosoughi K, Ichkhanian Y, Benias P, Miller L, Aadam AA, Triggs JR, Law R, Hasler W, Bowers N, Chaves D, Ponte-Neto AM, Draganov P, Yang D, El Halabi M, Sanaei O, Brewer Gutierrez OI, Bulat RS, Pandolfino J, Khashab M. Gastric per-oral endoscopic myotomy (G-POEM) for refractory gastroparesis: results from an international prospective trial. Gut. 2022 Jan;71(1):25-33. doi: 10.1136/gutjnl-2020-322756. Epub 2021 Mar 19. PMID 33741641